CLINICAL TRIAL: NCT04204980
Title: Desensitization in Kidney Allograft Recipients Before Transplantation Using Daratumumab
Brief Title: Desensitization in Kidney Allograft Using Daratumumab
Acronym: DARDAR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APHP190500
Record Dates: First submitted 2019-12-09; First posted 2019-12-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2023-02

CONDITIONS: Allosensitization; Kidney Transplant Rejection; Antibody-mediated Rejection
Keywords: Allosensitization; Kidney Transplantation

STUDY DESIGN:
Intervention Model Description: * Step I: dose-escalation 3 patients treated weekly during four weeks with 4 mg/kg of daratumumab, then 3 patients treated weekly during four weeks with 8 mg/kg of daratumumab, then 3 patients treated weekly four weeks with 16 mg/kg of daratumumab
  * Step II: expansion cohort to 13 patients (with 10 new patients included and the last 3 patients from the step I) with eight weekly doses of 16 mg/kg daratumumabProvide
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation and full dose (Experimental): Step I: dose-escalation 3 patients treated weekly during four weeks with 4 mg/kg of daratumumab, then 3 patients treated weekly during four weeks with 8 mg/kg of daratumumab, then 3 patients treated weekly four weeks with 16 mg/kg of daratumumab
  Step II: expansion cohort to 13 patients (with 10 new patients included and the last 3 patients from the step I) with eight weekly doses of 16 mg/kg daratumumab
  Interventions: Drug: Daratumumab dose escalation; Drug: Daratumumab full dose

INTERVENTIONS:
Drug: Daratumumab dose escalation — - Step I: dose-escalation 3 patients treated weekly during four weeks with 4 mg/kg of daratumumab, then 3 patients treated weekly during four weeks with 8 mg/kg of daratumumab, then 3 patients treated weekly four weeks with 16 mg/kg of daratumumab
Drug: Daratumumab full dose — - Step II: expansion cohort to 13 patients (with 10 new patients included and the last 3 patients from the step I) with eight weekly doses of 16 mg/kg daratumumab

SUMMARY:
Patients highly allosensitized against HLA antigen awaiting for a kidney transplant have less compatible transplants to them, increasing their waitlist time and mortality. Current desensitization strategies need to be improved with a high remaining acute rejection rate in this population and a substantial survival benefit which is not uniformly reported in the literature. The investigators propose to use daratumumab, a human IgG1 (Immunoglobulin Gamma-1) monoclonal antibody directed against the CD38 molecule (cluster of differentiation 38) witch induce response in refractory multiple myeloma by depleting plasma cells, as a new agent of desensitization. The study will address the hypothesis that daratumumab can lead to a significant decrease in calculated panel reactive antibodies by elimination of anti-HLA antibodies-producing plasma cells and facilitate the access to transplantation with a safety profile in highly sensitized patients registered in our kidney transplantation center.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years awaiting a kidney allograft transplantation
* Registration on the French National kidney allograft waiting-list for at least three years
* cPRA ≥ 95% for at least three years
* COVID-19 vaccination using Pfizer BioNtech vaccine for: Patients who have never been infected with COVID-19, inclusion at least one month after the third dose OR Patients previously infected with COVID-19 proved with PCR or serology, inclusion at least one month after the second injection of Pfizer BioNtech vaccine.
* Effective contraception up to three months after the end of treatment
* Informed consent obtained in accordance with local regulations;
* Affiliation to a social security regime.

Exclusion Criteria:

* Refusal of COVID-19 vaccination using Pfizer BioNtech vaccine
* Hypersensitivity to daratumumab or to any of the excipients),
* Known allergy to methylprednisolone and its excipients or to diphenhydramine and its excipients or to acetaminophen and its excipients or to valacyclovir and its excipients.
* Severe hepatocellular insufficiency
* Psychotic state not yet controlled by treatment
* Patient refusal
* Pregnant or breastfeeding woman or ineffective contraception
* Active neoplasia
* Active infection
* Active HBV infection, including HBsAg positive at screening
* Participation in another interventional study involving human participants or being in the exclusion period at the end of a previous study involving human participants
* Persons deprived of their liberty by judicial or administrative decision,
* Persons under legal protection/safeguard of justice,
* Patients under duress psychiatric care,
* Persons admitted to a health or social institution
* Patient on AME (state medical aid)
* Contraindication to kidney transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Serious adverse events (SAEs) and adverse event (AEs) related and unrelated to the treatment during the dose-escalation step | up to 21 months
Intra-patient variation of cPRA after daratumumab treatment | Baseline (Day 0) and at six months after daratumumab treatment

SECONDARY OUTCOMES:
Patient survival within one year after inclusion | Baseline (Day 0) and at six months after daratumumab treatment
Intra-patient variation of sum of mean fluorescence intensity (MFI) of anti-HLA antibodies | Baseline (Day 0) and at one month, three months, six months and 12 months after daratumumab treatment.Baseline (Day 0) and at one, three, six and 12 months after daratumumab treatment.
Intra-patient variation of cPRA (calculated panel reactive antibodies) after daratumumab treatment | Baseline (Day 0) and at one month, three months and 12 months after daratumumab treatment.
  PRA will be calculated on serum, analyzed with Luminex single antigen assays
Percentage of patients engrafted | At six months and 12 months after inclusion
Variation of immunoglobulin's blood titers | At baseline (Day 0), three months, six months and 12 months after daratumumab treatment
Intra-patient variation of ABO antibody titers | At baseline (Day 0), three months, six months and 12 months after daratumumab treatment
  ABO antibody titration will be performed by flow cytometry
Incidence of invasive infections | 6 months and on year after inclusion
Incidence of opportunistic infections | 6 months and one year after inclusion
Absolute number of Blood plasma cell | At baseline (Day 0), one month, three months , six months and 12 months after daratumumab treatment
Percentage of Blood plasma cell | At baseline (Day 0), one month, three months , six months and 12 months after daratumumab treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marie Matignon, MD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION